CLINICAL TRIAL: NCT06428487
Title: Phase II,Open-label, Non-randomized Study of Neoadjuvant Prolgolimab Monotherapy in Patients With Locally Advanced Colorectal Cancer With Microsatellite Instability (MSI)/Mismatch Repair (dMMR) Deficiency
Brief Title: Neoadjuvant Prolgolimab Monotherapy in Locally Advanced MMR-deficient Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Mikhail Fedyanin, Professor, Blokhin's Russian Cancer Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 125
Record Dates: First submitted 2024-03-05; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; immune checkpoint inhibitors; microsatellite instability
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolgolimab monotherapy (Experimental): The patients will be treated with prolgolimab 1 mg/kg every 2 weeks during 6 months (12 cycles) until surgery
  Interventions: Drug: Prolgolimab

INTERVENTIONS:
Drug: Prolgolimab — Prolgolimab infusions 1 mg/kg

SUMMARY:
In this phase II study patients with stage II-III MSI/dMMR colorectal adenocarcinoma with no signs of distant metastases will be treated with immunotherapy (prolgolimab). The duration of treatment is 6 months (12 cycles)

DETAILED DESCRIPTION:
In this open-label phase II non-randomized study the investigators will enroll 30 patients with stage II-III MSI/dMMR colorectal cancer to receive anti-PD1 inhibitor prolgolimab.

Patients will be treated with 12 cycles (6 months) of prolgolimab 1 mg/kg every 2 weeks until surgery.

ELIGIBILITY:
Inclusion Criteria:

* Availability of voluntarily signed informed consent from the patient
* Histologically confirmed adenocarcinoma of the colon or rectum;
* Locally advanced tumor - cT3-4N0-2M0 according to CT for tumors of the colon and sigmoid colon; cT3 with a depth of tissue invasion ≥5mm (cT2N0 and higher for lower ampullary cancer) or T4 or involvement of the lateral resection margins according to MRI for rectal cancer;
* Presence of MSI/dMMR in the tumor;
* ECOG 0-2;
* No contraindications to surgical treatment of malignancy

Exclusion Criteria:

* Previous therapy with the inclusion of monoclonal antibodies - anti-PD1, anti-PD-L1, anti PD-L2, anti-CTLA4 antibodies and other immunotherapy drugs
* The presence of any other malignant tumor, with the exception of radically treated basal cell carcinoma, cervical cancer in situ, currently or within 5 years before inclusion in the study
* Pregnant and lactating women, as well as planning pregnancy during the period of therapy in a clinical trial and 6 months after the end of therapy
* Patients with preserved reproductive potential who refuse to use adequate methods of contraception throughout the study and 6 months after the end of therapy or who agree to abstain from heterosexual contact.
* Previous systemic therapy with immunosuppressive drugs (including, but not limited to: prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide and TNF [tumor necrosis factor] antagonists) within 4 weeks before signing the informed consent form, or the need to use immunosuppressive therapy in during the first year of the study.
* The use of systemic glucocorticosteroids (GCS) in replacement doses (for example, in a dose equivalent to 10 mg of prednisolone per day or less), short-term use of systemic GCS (≤7 days), inhaled and topical GCS are allowed.
* Active, known or suspected autoimmune diseases (patients with type 1 diabetes mellitus and hypothyroidism requiring only hormone replacement therapy, as well as autoimmune diseases with only skin manifestations [for example, vitiligo, alopecia or psoriasis without symptoms of psoriatic arthritis] are allowed to participate), that do not require systemic therapy);
* Patients with HIV infection, active hepatitis B, active hepatitis C.
* Life expectancy less than 6 months.
* The presence of a disease or condition that, in the opinion of the investigator, prevents the patient from participating in the study.
* Complicated course of the primary tumor, requiring urgent surgical intervention.
* Previously performed radiation or chemotherapy for colorectal cancer, with the exception of cases of metachronous tumors over 5 years ago;
* Persistence, progression or recurrence of the underlying disease or the presence of distant metastases
* Conditions limiting the patient's ability to comply with the requirements of the protocol (in the opinion of the investigator);
* Vaccination with live vaccines within 28 days before randomization;
* Participation in other interventional clinical trials less than 30 days before randomization (except in cases of dropout before the introduction of study therapy) and while participating in an ongoing clinical trial;
* Significant adverse events from previous therapy, with the exception of chronic and/or irreversible events that cannot influence the assessment of the safety of the study therapy (for example, alopecia);
* Hypersensitivity or allergic reactions to the administration of drugs manufactured using Chinese hamster ovary cells, severe allergic reactions, anaphylaxis or other hypersensitivity reactions to chimeric or humanized antibodies, prolgolimab or any of the components of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | up to 8 months
  Absence of malignant cells on the specimen of colon/rectal resection in patients who were previously treated with neoadjuvant immunotherapy

SECONDARY OUTCOMES:
Durable complete clinical response rate (DRR) | up to 12 months
  a continuous response [complete or partial objective response] beginning within 6 months of treatment and lasting ≥6 months
Progression-free survival (PFS) | 12 months
  Time from initiation of treatment to the occurrence of disease progression or death.
Overall survival (OS) | 12 months
  Time from initiation of treatment to death.
Objective response rate (ORR) | up to 8 months
  percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)
R0 resection rate | up to 8 months
  Rate of R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed
Major pathologic response (MPR) | up to 8 months
  Rate of pathologic response TRG 1-2
Incidence of Treatment-Related Adverse Events as assessed by investigator | up to 6 months
  Incidence of Adverse Events assessed according to CTCAE version 5

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin NMRCO, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuznetsova O, Zagidullina A, Drobot N, Prokopiev A, Ivanov M, Fedyanin M, Mamedli Z, Aliev V, Polynovsky A, Dzhumabaev K, Aniskin A, Stroganova A, Karasev I, Tryakin A. Neoadjuvant Immunotherapy With Prolgolimab in Patients With Locally Advanced Microsatellite Instability/Defective Mismatch Repair Colorectal Cancer. JCO Precis Oncol. 2025 Dec;9:e2500602. doi: 10.1200/PO-25-00602. Epub 2025 Dec 10. PMID 41370727